CLINICAL TRIAL: NCT06834139
Title: Efficacy and Safety of the "Neo Pill" Device in Terms of Keeping Oral Hygiene and Health in Patients with Fixed Orthodontic Appliance
Brief Title: Efficacy and Safety of the "Neo Pill" Device for Keeping Oral Hygiene in Patients with Fixed Orthodontic Appliance
Acronym: NEOPILL
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Kragujevac (Other)
Responsible Party: Principal Investigator, Marko Milosavljević, Associated Professor, University of Kragujevac
Other Study IDs: 01-3909
Record Dates: First submitted 2025-02-10; First posted 2025-02-19 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Oral Hygiene

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Neo Pill group: The Neo Pill group include patients with fixed orthodontic appliance who will use Neo Pill device for improving oral hygiene.
- Control group: The Control group will include patients with fixed orthodontic appliance who will not use Neo Pill device, but will keep oral hygiene in conventional way (toothbrush, etc.)

SUMMARY:
Background: Orthodontic appliances interfere with oral hygiene and contribute to plaque retention, gingival inflammation and demineralization of enamel. Current techniques for keeping oral hygiene (teeth brushing, rinsing oral cavity with 0.12% chlorhexidine, dental floss, interdental brush, Miswak) are not sufficiently effective (1). Up to 78% of patients do not follow instructions to keep oral hygiene with current methods which require discipline and effort (2). There is great need for some simple medical device to keep oral hygiene in an effective, safe and easy-to-use way.

Objective: To evaluate efficacy and safety of NeoPill electrolysis device for keeping oral hygiene in patients with fixed orthodontic appliances.

Hypotheses: (1) NeoPill electrolysis device in addition to standard oral hygiene techniques improves values of oral health indices (gingival bleeding index, papillary bleeding index, plaque index, and ortho-plaque index) and is associated with fewer white spots on enamel during and after 6 months of use in comparison to standard oral hygiene techniques only; (2) the adverse event rates in patients using the NeoPill electrolysis device and in patients keeping oral hygiene only with standard techniques is not significantly different; (3) quality of life in patients using the NeoPill electrolysis device is higher than in patients keeping oral hygiene only with standard techniques.

Methods: The study is designed as prospective cohort investigation. Primary outcomes of the study are: the Turesky Modified Quigley Hein Plaque Index (TQHPI) for both anterior and posterior teeth Gingival Inflammation Score (GIS) for both anterior and posterior teeth, Papillary bleeding index (PBI), Ortho-Plaque Index (OPI), number of white spots on enamel, and safety (incidence of adverse events). Secondary outcomes are quality of life and overall costs of keeping oral hygiene. Main independent variable in the study is administration of the NeoPill electrolysis device produced by start-up innovative company Laviefarm, Belgrade, Serbia. The device causes detachment of bacteria from fixed orthodontic appliances and teeth, which are then washed out with mouth rinse, and swallowed or spitted out.

Implications and significance: If proved effecive and safe, the NeoPill electrolysis device will make major contribution to improvement of oral hygiene in patients with fixed orthodontic appliances.

DETAILED DESCRIPTION:
BACKGROUND AND SIGNIFICANCE Fixed prosthetic appliances can pose a challenge to maintaining oral hygiene. The placement of fixed orthodontic appliances, for example, can compromise the patient's oral environment through the presence of additional surfaces and impeding oral hygiene procedures, which can affect the oral microbiota balance. Rough and irregular margins on the fixed prosthetic constructions can also result in microorganisms' attachment, which can worsen oral hygiene conditions and cause gingivitis and further periodontitis .

Oral hygiene practices include brushing with fluoride toothpaste, flossing, using mouthwash, and avoiding sugary foods and drinks. Brushing should be done at least twice a day, using a soft-bristled toothbrush and a 45-degree angle to the gumline. Flossing should be done daily, using a floss threader or an interdental brush to clean between the teeth and under the wires. Mouthwash can help reduce plaque and inflammation, but should not replace brushing and flossing. Sugary foods and drinks can increase the risk of tooth decay and enamel demineralization.

Oral hygiene status can be assessed by using different indices, such as the Orthodontic Plaque Index, the Gingival Index, and the Bleeding Index. These indices measure the amount of plaque, inflammation, and bleeding in the gingival tissues around the orthodontic appliances. The oral hygiene status can also be visualized by using disclosing tablets or toothpaste, which stain the plaque and show where it needs to be removed.

Oral hygiene in patients with fixed orthodontic appliances is not satisfactory in majority of cases. There is significantly higher frequency of signs of gingival inflammation and amount of dental plaque in patients with fixed orthodontic appliances. The pocket probing depth, total number of microorganisms and number of patients with positive findings of Prevotella intermedia and other periodontopathic anaerobes are increased after wearing fixed orthodontic apppliance. Prolonged treatment increases the risk of plaque development around orthodontic brackets and bands. This can further lead to heightened risk for caries development and higher possibility of white spot lesions development around fixed orthodontic brackets. Among these devices, stainless steel lingual retainers, plain or braided, have much less periodontal complications then glass-fibre reinforced retainers, but they still require intensive dental hygiene if gingival inglammation, dental plaque and white spots at enamel are to be avoided.

There is great need for some simple medical device to keep oral hygiene in an effective, safe and easy-to-use way. Recently an innovation in this field has been made, and NeoPill electrolysis device was developed, which causes detachment of bacteria from the fixed appliance and their rapid elimination. Although the device was approved for sale and human use in Serbia, for wider use it is necessary to prove its efficacy and safety in clinical studies, what is exactly the intention of this project. If proved to be safe and effective, this device could revolutionize oral hygiene practices and help preventing developing of periodontal disease and carries.

LITERATURE REVIEW:

The human oral cavity provides a habitat for oral microbial communities, including bacteria, archaea, fungi, viruses, and protozoa. The complexity of its anatomical structure, its connectivity to the outside, and its moist environment contribute to the complexity and ecological site specificity of the microbiome colonized therein. The dysbiotic state, in which the microbial composition is altered and the microecological balance between host and microorganisms is disturbed, can lead to oral and even systemic diseases. There is specificity of the microbiota at different niches in the oral cavity, and various communities of the oral microbiome exist: the mycobiome, the bacteriome, and the virome within oral biofilms . Although there is no definitive list of pathogenic bacteria in oral microbioma, some bacteria are known to be associated with oral diseases. For example, Streptococcus mutans is known to cause dental caries. Porphyromonas gingivalis and Treponema denticola are associated with periodontitis, and Prevotella intermedia is associated with gingivitis.

Fixed orthodontic appliances can affect the oral environment and microbiome by creating conditions that favor plaque accumulation and biofilm formation. The fixed orthodontic treatment also impedes oral hygiene procedures. This can lead to increased levels of microorganisms in saliva and dental plaque, especially anaerobic and facultative anaerobes, such as Streptococcus mutans, Fusobacterium, Treponema, Porphyromonas, Tannerella, Campylobacter, and Prevotella. The appliances can act as anchors for biofilm and plaque formation, leading to an accumulation of bacteria and other microorganisms in amounts unfavorable for maintaining a healthy equilibrium. This can cause dysbiosis, which manifests clinically as increased enamel demineralization, dental caries, and periodontal disease. The changes in the oral microbiome induced by fixed orthodontic appliances are dynamic and may be influenced by the type of appliance, the surface properties of the biomaterials, the duration of treatment, and the oral hygiene practices of the patients. Maintaining proper oral hygiene and using fluoride mouthwash are important factors to mitigate the harmful effects of dysbiosis and prevent secondary infections.

Efficacy of classic methods of keeping oral hygiene is decreased in patients with fixed orthodontic appliances. The efficacy of three types of manual toothbrushes (Cross action, Flat trim, and orthodontic type) in terms of plaque removal in patients undergoing fixed orthodontic treatment was investigated in a three-treatment, three-period crossover clinical trial with a single brushing exercise. The primary outcome measure was the difference in the plaque scores (baseline minus post-brushing) at each study period, as determined by the Turesky-Modified Quigley-Hein Plaque Index. The results showed that the Flat trim toothbrush was significantly better at reducing plaque than the Orthodontic type and Cross action types. No significant differences were found between the Orthodontic type and Cross action types.

Another study compared the cleansing efficacy of an oral irrigator with that of dental flossing in patients with fixed braces after 4 weeks of home-use. The study concluded that dental floss is more effective than oral irrigators in removing plaque and reducing gingival bleeding in easily accessible regions. However, in posterior regions, where patients struggled with the application of dental floss, the oral irrigator showed similar results. A study published in the European Journal of Orthodontics found that interdental brushes are effective in removing plaque and reducing gingival bleeding in patients undergoing fixed orthodontic therapy. The study concluded that the percentage of patients with excellent oral hygiene increased from 19% to 41% after using interdental brushes.

A systematic review of clinical trials evaluated the effect of chlorhexidine mouth rinse on plaque, gingival bleeding and gingival pocket depth in orthodontic patients with fixed appliances. The study concluded that adding chlorhexidine mouth rinse to the daily oral hygiene regimen reduces plaque and gingivitis development and is effective in improving the appearance of gingiva in orthodontic patients. Another study evaluated the effect of 40% chlorhexidine varnish on gingival health in patients with fixed orthodontic appliances and increased gingival volume. The varnish was applied on the vestibular area of the upper premolars and first molar crowns. The use of 40% CHX varnish decreased the gingival overgrowth in patients undergoing orthodontic treatment. Further studies are necessary to set the action time and frequency of application. Chlorhexidine varnish also decreased the level of mutans streptococcus and lactobacillus colonies, and the development of white spot lesions in patients with fixed orthodontic appliances, when tested in a study on 32 volunteers. The varnish was applied monthly around the brackets and tubes.

A clinical study evaluated the efficacy of Miswak in comparison to a toothbrush in reducing dental biofilm and gingivitis in patients with fixed orthodontic appliances. The study concluded that Miswak is effective in reducing dental biofilm and gingivitis. Miswak is a natural toothbrush made from the twigs of the Salvadora persica tree, which has been used for centuries in traditional oral hygiene practices. Miswak contains natural antimicrobial compounds such as tannins, flavonoids, and alkaloids that can help reduce the levels of microorganisms in the oral cavity.

However, fixed orthodontic appliances patients suffer limitations on the effective control of biofilm by mechanical methods, bringing the need of a coadjutant in the control of inflammation and oral health improvement. Additionally, compliance of the patients to recommended schedule and techniques of teeth brushing, interedental brushing, dental floss, Miswak or mouthrinsing could be problematic. A study by Buthelezi et al found that most patients undergoing fixed orthodontic treatment had satisfactory oral hygiene status and habits. The majority of patients avoided sticky foods, used mouthwash, flossed daily, and brushed twice daily. However, 82% of them consumed sugar-containing drinks. The study also found that younger patients had better gingival health than older patients. Another study assessed the knowledge, attitude, and practice of patients towards orthodontic treatment. This study concluded that the orthodontic patients possess good knowledge about their treatment; however, their attitude and orthodontic related practices need to be improved. In general, females and those with tertiary education fared better for all three domains. It was also found that it is necessary to practice a structured follow-up communication after orthodontic appliance application in order to improve oral hygiene compliance.

Specialized devices for improving oral hygiene using physical forces other than mechanical are rarely used. As a result of literature search only one device was found, called Photomedics BlueLight. This device has been developed and designed to reduce the number of potentially pathogenic oral bacteria that can cause gum disease and bad breath and are linked to cardiovascular disease, stroke, premature birth, and low birth weight. The device uses blue light of the appropriate wavelength and intensity to target and kill only the harmful, disease-causing bacteria while allowing helpful bacteria to thrive and rebalance the oral microbiome .

In summary, fixed orhtodontic appliances are associated with increased number of pathogenic bacteria and formation of biofilm, that causes gingivitis and white spots on enamel, a precursor of dental caries. Although mechanical means for keeping oral hygiene are effective in prevention of gingivitis and white spots if regularly and appropriately applied, it is difficult to achieve full protection in everyday life due to incomplete patient compliance and limited access to posterior teeth. There is great unmet need to develop innovative devices for keeping oral hygiene in patients with fixed orthodontic appliances, that would be effective, easy-to-use and safe.

RESEARCH DESIGN AND METHODS STUDY DESIGN: Prospective Cohort Study PRIMARY OBJECTIVES

* To investigate effectiveness of NeoPill electrolysis device for keeping hygiene of oral cavity in patients with fixed orthodontic appliances
* To investigate safety and tolerability of NeoPill electrolysis device for keeping hygiene of oral cavity in patients with fixed orthodontic appliances

SECONDARY OBJECTIVES

* To investigate quality of life on a VAS scale when NeoPill electrolysis device is used for keeping hygiene of oral cavity in patients with fixed orthodontic appliances
* To investigate costs of NeoPill electrolysis device use for keeping hygiene of oral cavity in patients with fixed orthodontic appliances

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Fixed orthodontic appliance in place for at least 15 days
* Aged 18 years or above
* Good general health
* Permanent dentition
* Less than 5 mm of anterior crowding or spacing with adequate overjet and overbite
* Ability to maintain adequate oral hygiene
* Optimum dental health without immediate need for any allied dental procedure

Exclusion Criteria:

* Pregnancy, anticipated pregnancy, or breastfeeding
* Incarceration or institutionalized living
* Participation in another clinical study
* Life expectancy <4 months
* Patients with moderate to severe renal insufficiency (acute or chronic) with glomerular filtration rate of less than 30 ml/min
* Patients with active bronchospastic disorders
* Heart failure classes III and IV
* Active dental caries
* Active periodontal disease
* Chronic systemic diseases
* Using antibiotics within the last 30 days
* Skeletal anteroposterior discrepancies between the maxilla and the mandible (ANB equal or above 5 degrees)
* Centric relation-centric occlusion discrepancies greater than 3 mm
* Patients with pace-makers and other implanted devices that require stable supply by electric energy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with Fixed orthodontic appliance in place
Sampling Method: Non-Probability Sample
Enrollment: 143 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
1. The Turesky Modified Quigley Hein Plaque Index (TQHPI) for both anterior and posterior teeth | 6 months
  This is the scale (questionnaire), unit of measurement is the score of the scale.
2. Gingival Inflammation Score (GIS) for both anterior and posterior teeth | 6 months
  This is the scale (questionnaire), unit of measurement is the score of the scale.
Papillary bleeding index (PBI) | 6 months
  This is the scale (questionnaire), unit of measurement is the score of the scale.
Ortho plaque index | 6 months
  This is the scale (questionnaire), unit of measurement is the score of the scale.
Number of white spots on enamel | 6 months
  It is measured by direct observation of the teeth; the unit of measurement is number of white spots.
Safety (incidence of adverse events) | 6 months
  Adverse events are recorded by direct observation and interview with the patients. Unit of measurement is number of adverse events.

SECONDARY OUTCOMES:
Costs of treatment | 6 months
  Costs of treatment are measured by the multiplication of resource utilization figures with unit prices; units of measurement are RSD (Republic of Serbia Dinars)

CONTACTS AND LOCATIONS:
Overall Officials: Slobodan Janković, DSc, MD, Study Chair — University of Kragujevac, Faculty of Medical Sciences
Locations (1):
- University of Kragujevac, Faculty of Medical Sciences, Kragujevac, Serbia, Serbia

IPD SHARING:
Plan to Share IPD: No